CLINICAL TRIAL: NCT00336232
Title: Dietary and Non-dietary Components of Vitamin K Metabolism
Brief Title: Determinants of Vitamin K Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Sarah Booth, Senior Scientist, Tufts University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01DK069341 (NIH)
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Aging; Osteoporosis
Keywords: Vitamin K metabolism; Bone health; Metabolism
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin K; Vitamin K 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diet Intervention (Experimental): 28 day diet low vitamin K, 28 day diet high vitamin K
  Interventions: Drug: Vitamin K

INTERVENTIONS:
Drug: Vitamin K — phylloquinone (vitamin K1) 500 mcg daily in third month
  Other Names: phylloquinone

SUMMARY:
The purpose of this study is to learn how the body responds to different amounts of vitamin K in the diet in order to understand the roles that vitamin K may have in the body. We also need to determine if older adults need more or less vitamin K in their diet compared to younger adults in order to maintain normal body stores of vitamin K.

DETAILED DESCRIPTION:
Vitamin K has a role in bone health, but little is known about vitamin K metabolism in aging and in maintenance of bone mass. The limited understanding of vitamin K metabolism impedes the establishment of dietary recommendations for vitamin K, and the interpretation of results from clinical trials on vitamin K supplementation and bone health of women in a narrow age group. This study is the first to assess the role of dietary and other factors that influence the response to vitamin K status and bone turnover to vitamin K depletion and repletion in adults. This study also compares the absorption efficiency and body retention of vitamin K relative to current vitamin K status. Men and women [21 younger (18-40y) and 21 older (55+y)] will participate in a 62-d metabolic study, with a 5d run-in period, followed by a 28d dietary vitamin K restriction period (10 ug/d), and ending with a 28d dietary vitamin K supplementation period (500 ug/d). Coagulation times will be monitored during the dietary restriction period. Serial measurements of vitamin K status markers and of bone turnover markers will show the response of vitamin K to dietary manipulation for both age groups under identically controlled dietary conditions. Deuterium-labeled vitamin K in collards will be used to compare the absorption of vitamin K during a vitamin K-deplete state to that of a vitamin K-replete state. Vitamin K is transported in triglyceride-rich lipoproteins, which may vary among individuals due to differences in adiposity and lipid homeostasis. Therefore, measurement of body composition by Dual Energy X-Ray Absorptiometry (DXA) and plasma lipids will provide insight into the role of lipids in absorption and transport of vitamin K. The findings of this study are critical for the interpretation of the epidemiologic and clinical data used to determine the protective role vitamin K may have in chronic disease prevention.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* kidney, GI, or liver disease requiring treatment
* prescribed osteoporosis medications in the previous 3 months
* use of acid reducers more than twice per week
* blood clotting disorder and/or abnormal clotting time
* warfarin or anticoagulant use in the previous 12 months
* diabetes
* smoking
* hormone therapy in the previous 3 months
* oral contraceptive use in the previous 3 months; pregnancy
* strict vegetarian diet

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Booth, PhD, Principal Investigator — Tufts Medical Center
Locations (1):
- Jean Mayer United States Department of Agriculture Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Harrington DJ, Soper R, Edwards C, Savidge GF, Hodges SJ, Shearer MJ. Determination of the urinary aglycone metabolites of vitamin K by HPLC with redox-mode electrochemical detection. J Lipid Res. 2005 May;46(5):1053-60. doi: 10.1194/jlr.D400033-JLR200. Epub 2005 Feb 1. PMID 15722567
- [Background] Erkkila AT, Lichtenstein AH, Dolnikowski GG, Grusak MA, Jalbert SM, Aquino KA, Peterson JW, Booth SL. Plasma transport of vitamin K in men using deuterium-labeled collard greens. Metabolism. 2004 Feb;53(2):215-21. doi: 10.1016/j.metabol.2003.08.015. PMID 14767874
- [Background] Booth SL, Martini L, Peterson JW, Saltzman E, Dallal GE, Wood RJ. Dietary phylloquinone depletion and repletion in older women. J Nutr. 2003 Aug;133(8):2565-9. doi: 10.1093/jn/133.8.2565. PMID 12888638
- [Background] Booth SL, Lichtenstein AH, O'Brien-Morse M, McKeown NM, Wood RJ, Saltzman E, Gundberg CM. Effects of a hydrogenated form of vitamin K on bone formation and resorption. Am J Clin Nutr. 2001 Dec;74(6):783-90. doi: 10.1093/ajcn/74.6.783. PMID 11722960
- [Result] Traber MG, Leonard SW, Bobe G, Fu X, Saltzman E, Grusak MA, Booth SL. alpha-Tocopherol disappearance rates from plasma depend on lipid concentrations: studies using deuterium-labeled collard greens in younger and older adults. Am J Clin Nutr. 2015 Apr;101(4):752-9. doi: 10.3945/ajcn.114.100966. Epub 2015 Mar 4. PMID 25739929
- [Result] Truong JT, Fu X, Saltzman E, Al Rajabi A, Dallal GE, Gundberg CM, Booth SL. Age group and sex do not influence responses of vitamin K biomarkers to changes in dietary vitamin K. J Nutr. 2012 May;142(5):936-41. doi: 10.3945/jn.111.154807. Epub 2012 Mar 21. PMID 22437558
- [Derived] Ellis JL, Fu X, Al Rajabi A, Grusak MA, Shearer MJ, Naumova EN, Saltzman E, Barger K, Booth SL. Plasma Response to Deuterium-Labeled Vitamin K Intake Varies by TG Response, but Not Age or Vitamin K Status, in Older and Younger Adults. J Nutr. 2019 Jan 1;149(1):18-25. doi: 10.1093/jn/nxy216. PMID 30590596
- See also: Jean Mayer USDA Human Nutrition Research Center on Aging site — http://hnrc.tufts.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin K Diet Intervention: 5 day baseline vitamin K
  Vitamin K: phylloquinone (vitamin K1) 200 mcg daily
  28 day diet low vitamin K
  Vitamin K: phylloquinone (vitamin K1) approx. 10 mcg daily for 28 days
  treatment started day 6, completed day 33
  28 day diet high vitamin K
  Vitamin K: phylloquinone (vitamin K1) 500 mcg daily in third month
  treatment started day 34, ended day 61
Period: Baseline (200mcg Daily)
Arm/Group | Vitamin K Diet Intervention
Started | 59
Completed | 42
Not Completed | 17
Period: Low Vitamin K (10mcg Daily)
Arm/Group | Vitamin K Diet Intervention
Started | 42
Completed | 42
Not Completed | 0
Period: High Vitamin K (500mcg Daily)
Arm/Group | Vitamin K Diet Intervention
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Diet Intervention: 5 day baseline vitamin K
  Vitamin K: phylloquinone (vitamin K1) 200 mcg daily
  28 day diet low vitamin K
  Vitamin K: phylloquinone (vitamin K1) approx. 10 mcg daily for 28 days
  treatment started day 6, completed day 33
  28 day diet high vitamin K
  Vitamin K: phylloquinone (vitamin K1) 500 mcg daily in third month
  treatment started day 34, ended day 61
Arm/Group | Diet Intervention
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 32
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 42
Plasma phylloquinone (nmol/L) [Mean (Standard Deviation); unit: nmol/L] | 0.8 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Phylloquinone
Description: Plasma phylloquinone in response to phylloquinone depletion and repletion
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Diet Intervention
Number analyzed (Participants) | 42
nmol/L
  low vitamin K | 0.3 (0.6)
  high vitamin K | 2.3 (1.4)

ADVERSE EVENTS:
Time Frame: duration of study, up to 62 days
Arm/Group | Diet Intervention
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 3/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diet Intervention (N=42)
High blood pressure (Blood and lymphatic system disorders) | 1 (1) — not related to intervention
History of blood clotting (Blood and lymphatic system disorders) | 1 (1) — ineligible for study enrollment
Facial swelling (General disorders) | 1 (1) — not related to intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No